CLINICAL TRIAL: NCT00882973
Title: Trial to Determine the Maximum Tolerated Dose of Genexol-PM Plus Gemcitabine and Evaluate Efficacy and Safety of Genexol-PM Regimens in Subjects With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: GPMPC202
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — genexol-PM

ARMS (3):
- Cohort 1 (Experimental): Genexol-PM 220 mg/m2 + Gemcitabine 1,250 mg/m2
  Interventions: Drug: Genexol-PM
- Cohort 2 (Experimental): Genexol-PM 260 mg/m2 + Gemcitabine 1,250 mg/m2
  Interventions: Drug: Genexol-PM
- Cohort 3 (Experimental): Genexol-PM 300 mg/m2 + Gemcitabine 1,250 mg/m2
  Interventions: Drug: Genexol-PM

INTERVENTIONS:
Drug: Genexol-PM — Cremophor EL-free polymeric micelle of paclitaxel

SUMMARY:
This is a phase I/II trial to determine the maximum tolerated dose and recommended phase II dose of the combination therapy with Genexol-PM and gemcitabine (hereafter Genexol-PM plus gemcitabine) and to evaluate the efficacy and safety of Genexol-PM regimens (monotherapy and combination with gemcitabine) and gemcitabine monotherapy in subjects with locally advanced or metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who aged 18 years or older
2. Subjects whose written informed consent was obtained complying with the local regulatory requirements prior to their participation in the trial
3. Subjects who have histologically or cytologically confirmed unresectable or metastatic epithelial cancer of the exocrine pancreas. High-quality contrast-enhanced CT scanning is required to evaluate resectability. Measurable disease is not required.
4. Subjects with no other malignancy diagnosed within past five years except for:

   * Cured non-melanoma skin cancer
   * Cured cervical intraepithelial neoplasia (CIN)
   * Cured In-situ cervical cancer (CIS)
5. Subjects who are ECOG performance status of ≤ 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2009-08 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) of the combination therapy with Genexol-PM and gemcitabine | 1 year
The recommended phase II dose of the combination therapy with Genexol-PM and gemcitabine | 1 year

SECONDARY OUTCOMES:
Objective response rate (complete response (CR) + partial response (PR)) | 1 year
Time to tumor progression | 1 year
Progression free survival | 1 year
Safety profiles | 1 year